CLINICAL TRIAL: NCT06804447
Title: Pencil Beam Scanning Proton Beam Radiotherapy for the Management of Abdominal Neuroblastoma - an Evaluative Commissioning in Protons (ECIP) Study
Brief Title: Pencil Beam Scanning Proton Beam Radiotherapy for the Management of Abdominal Neuroblastoma
Acronym: SUPERMAN
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Christie NHS Foundation Trust (Other)
Collaborators: University College London Hospitals (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CFTSp218 (03); NPBT3211 (Other Grant/Funding Number: NHS England)
Record Dates: First submitted 2025-01-08; First posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Abdominal Neuroblastoma
Keywords: Proton Beam Therapy; Abdominal Neuroblastoma; Evaluative Commissioning
MeSH Terms: interventions — Proton Therapy

STUDY DESIGN:
Intervention Model Description: SUPERMAN is a multicentre prospective study assessing the feasibility of using an algorithm based on pre-defined clinical characteristics to appropriately select patients with abdominal or abdominal-pelvic neuroblastoma for PBT treatment. This study will also assess delivered dosimetry of PBT plans with adaptive treatment strategies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Radiotherapy (Other): Proton Beam Radiotherapy (PBT) or Intensity Modulated Radiotherapy (IMRT)
  Interventions: Radiation: Proton Beam Therapy

INTERVENTIONS:
Radiation: Proton Beam Therapy — Proton Beam Therapy

SUMMARY:
Proton Beam Therapy (PBT) and Evaluative Commissioning in Protons (ECIP):

PBT is an advanced radiotherapy technique. There are two National Health Service (NHS) PBT treatment centres in the United Kingdom, in Manchester and London. The NHS is committed to ensuring the best use of this limited resource by investigating which patients will benefit from PBT. ECIP is a programme of studies exploring the role of PBT in different types of cancer funded by NHS England. ECIP studies are not randomised, eligible patients will be offered PBT. Any eligible UK patient can be referred, and accommodation is available for patients who don't live close to a PBT centre. The main benefit of PBT, compared with standard photon radiotherapy, is predicted reduction in radiation dose to surrounding healthy tissues. With photon radiotherapy, some radiation passes beyond the target area, affecting healthy tissues and causing side-effects. With PBT, the radiation dose stops within the target area, causing less damage to surrounding tissues, and limiting side effects.

SUPERMAN:

SUPERMAN is a study within the ECIP programme. It is sometimes not entirely clear whether PBT or photon radiotherapy is better for the treatment of a patient with abdominal neuroblastoma. The aim of SUPERMAN is to choose the best radiotherapy technique and to better understand how to monitor and adapt PBT for these patients.

DETAILED DESCRIPTION:
Introduction:

Neuroblastoma is a rare childhood cancer, occurring in about 100 children in the UK each year. Most arise from nerves in the retroperitoneum - this is an area at the back of the abdomen, behind the stomach and bowel. There are many important structures in the retroperitoneum including the kidneys, adrenal glands, and parts of large blood vessels.

The treatment of neuroblastoma can include surgery, chemotherapy and radiotherapy. Radiotherapy is typically delivered after chemotherapy and surgery, depending on the response to previous treatments. Its aim is to improve local control and overall survival. The dose and schedule of radiotherapy is currently being investigated in a randomised Phase III pan-European trial called SIOPEN-HR-NBL2 (European Society for Paediatic Oncology High-Risk Neuroblastoma 2 trial). It is important to note that any patients involved in SUPERMAN will also be able to participate in any other radiotherapy study, including SIOPEN-HR-NBL2.

How advanced radiotherapy techniques can reduce treatment related side effects:

Typically, patients are diagnosed with neuroblastoma at a very young age, usually under 5 years old. There is a risk of late side-effects following radiation treatment, including secondary cancers. The risk of late-effects, and their severity, may be worse if patients already have health problems, such as problems with kidneys. Kidney problems may be due to the cancer itself or prior treatments. Therefore, particularly for patients most at risk, it is critical to reduce radiotherapy related side effects as much as possible.

In recent years, advances in photon (x-ray) radiotherapy, have improved the accuracy of treatment and reduced high dose radiation to nearby healthy tissues, reducing treatment related side-effects. However, these techniques increase the amount of normal tissue receiving low doses of radiation, and there are concerns about the increased risk of secondary malignancy. This is particularly important in the paediatric population. There will be no increased risk of secondary malignancy from participation in the study.

Proton Beam Therapy (PBT) is a different type of radiotherapy, in which charged particles (protons), rather than photons, are used to deliver treatment. It can potentially reduce the irradiation of nearby healthy tissues even further.

The use of PBT, and the subsequent improved radiation spread in the body, is associated with reduced radiotherapy side effects. The risk of developing radiation induced secondary malignancies for patients with abdominal neuroblastoma has also been estimated to be lower with PBT compared to photon radiotherapy.

The challenges of proton beam therapy and rationale for the study:

Despite the clear potential advantages of PBT, it may not be the best technique for all patients. SUPERMAN aims to address the questions around the decision-making processes for patient selection where the benefits of PBT are uncertain.

PBT treatments are more sensitive to changes in the body. If the body shape changes (e.g. the patient changes weight), or if there are changes inside the body (e.g. as organs move during respiration, or the bowel contains more or less gas than planned for), this could result in the radiotherapy going to the wrong place. Either too much or too little radiotherapy may treat the target region, or too much may be delivered to healthy tissues. The impact of these changes is different for each patient. In SUPERMAN, detailed monitoring of internal motion during treatment will allow us to monitor and estimate its importance for each patient - helping us to tailor treatment accordingly.

These challenges with PBT treatment delivery have led to mixed opinions amongst international experts as to whether there is a benefit with PBT for all neuroblastoma patients. Some groups have retrospectively published their limited experience of using PBT for neuroblastoma, but none have adequately reported on the assessment and management of the relevant changes in the body during treatment. It is therefore unclear from these studies if all neuroblastoma patients can safely be treated with PBT compared to photon delivery methods. A virtual comparative double planning study of PBT versus proton radiotherapy on twenty abdominal neuroblastoma patients has demonstrated that, although most cases will receive a superior treatment plan with PBT, a small proportion would be better served with photon techniques.

Currently policy and aims of the study:

PBT is currently commissioned for all paediatric and teenage young adult patients with abdominal neuroblastoma for whom there is thought to be an advantage. However, knowing who will benefit is not always clear. In some cases, a significant amount of planning needs to be done before a decision can be reached. This leads to uncertainty for everyone, including the patient. We estimate that roughly 10-15% of patients may be better off receiving advanced photon radiotherapy. A decision tool to guide decision making will help clinicians, support patients and improve treatment efficacy and resource use.

Several characteristics are thought to be important when deciding whether PBT or photons would be best for patients. These include the location and size of the tumour before surgery. By studying these factors in detail within SUPERMAN, it is hoped they could be accurately used within a decision tool to decide a patient's best treatment without delay.

Thus, the primary aim of SUPERMAN is to create an easy guide to support the decision-making between PBT and photon techniques, reducing uncertainty and improving treatment efficiency.

SUPERMAN is a multicentre prospective study assessing the feasibility of using an algorithm based on pre-defined clinical characteristics to select patients appropriately with abdominal or abdominal-pelvic neuroblastoma for PBT treatment. This study will also assess delivered dosimetry of PBT plans with adaptive treatment strategies.

Patient identification and referral will follow and leverage the standard pathways and processes for routinely commissioned indications in protons. Patients can potentially be identified at any centre treating this group of patients and referred to the study/PBT centres for consideration for study participation and radiotherapy treatment.

There will be two parts to this study - Technique Selection (Part A) and PBT Treatment Deliverability (Part B). Patients can be enrolled onto either one or both parts of this study.

Part A: Technique Selection

At the time of PBT referral, patients will be stratified into two groups:

* Proton clear benefit - Patients in this group will be treated with protons via the routine commissioning pathway. Patient criteria for this group is based on anatomical location.
* Proton potential benefit - Patients in this group will be offered enrolment onto Part A of the ECIP study. A "Technique Selection Algorithm" will be used as a process to determine the best modality (PBT or photon radiotherapy) for treatment delivery. Factors such as pre-radiation organ function (in particular kidneys), balance between target volume dose coverage versus sparing of organs at risk (OAR) and robustness of the PBT plan will be carefully considered in this algorithm. Double planning may be required to assist the decision-making process.

Part B: PBT Treatment Deliverability All patients who have PBT technique selected for treatment delivery either on the routine commissioning pathway or Part A should be offered enrolment into Part B of the study. This part of the study will entail detailed monitoring and dosimetric assessment of patients receiving PBT.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with histologically confirmed abdominal or abdominal-pelvic neuroblastoma who are eligible and fit for radical radiotherapy.
* Written informed consent from patient, parent or guardian - this includes consent for the minimum baseline, treatment and follow up assessments; and for their data to be stored and used for research, within the appropriate Proton Clinical Outcomes Units and NHS Proton Registry.
* Patients registered female at birth of childbearing potential agree to use effective contraception between the planning Computed Tomography (CT) scan and the end of treatment.

Exclusion Criteria:

* Pregnant patient

Min Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2030-03-01 (Estimated); Study Completion 2030-03-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of decision regarding radiotherapy technique selection at three time points of the patient and radiotherapy pathway | From date of first patient enrolment until the date of the last patient treatment (up to 36 months)
  Comparison of decision regarding radiotherapy technique selection (PBT vs IMRT) at three time points of the patient and radiotherapy pathway:
  1. Selection 1 - Proposed modality at time of referral - Pre-planning
  2. Selection 2 - Post planning
  3. Selection 3 - Post completion of radiotherapy

SECONDARY OUTCOMES:
Measure and compare dose to target volume of PBT versus IMRT plans. | From date of first patient enrolment until the date of the last patient treatment (up to 36 months)
  For patients who are dual planned, measure and compare dose to target volume, organs at risk and normal tissues of PBT versus IMRT plans (this is a descriptive endpoint).
Measure and compare dose to organs at risk of PBT versus IMRT plans. | From date of first patient enrolment until the date of the last patient treatment (up to 36 months)
  For patients who are dual planned, measure and compare dose to target volume, organs at risk and normal tissues of PBT versus IMRT plans (this is a descriptive endpoint).
Measure and compare dose to normal tissues of PBT versus IMRT plans. | From date of first patient enrolment until the date of the last patient treatment (up to 36 months)
  For patients who are dual planned, measure and compare dose to target volume, organs at risk and normal tissues of PBT versus IMRT plans (this is a descriptive endpoint).
Number of PBT re-plans and reasons (including delays) | From date of first patient enrolment until the date of the last patient treatment (up to 36 months)
  Number of PBT re-plans and reasons (including delays)
Number of patients requiring PBT to IMRT treatment modality conversions and the reasons for this. | From date of first patient enrolment until the date of the last patient treatment (up to 36 months)
  Number of patients requiring PBT to IMRT treatment modality conversions and the reasons for this.
Evaluation of on-treatment imaging | From date of first patient enrolment until the date of the last patient treatment (up to 36 months)
  Monitoring of PBT treatment deliverability, close monitoring of changes in anatomy and variable tissue heterogeneity during treatment is required to ensure that any required adaptive replans can be done within a timely fashion.
  Patients should have daily kV on board imaging and daily cone beam CT (CBCT) acquired for verification. If changes in anatomy is observed on CBCT, the impact on dosimetry on the current plan will need to be assessed. A traffic light system will be used to evaluate if dosimetric calculation is necessary.
Evaluation of on-treatment delivery data | From date of first patient enrolment until the date of the last patient treatment (up to 36 months)
  The methodology of evaluating on treatment imaging verification and clinical impact of dosimetric assessment during treatment has been described in the outcome measure above.
  The proportion of CBCTs graded green, amber and red will be recorded. The reasons for amber and red grading will be collected such as bowel gas changes or contour changes along with the attempted strategies applied to mitigate this.
  The reasons and proportion of patients who required replanning will be recorded and reported. The reasons and proportion of patients initially selected for PBT who required replanning for IMRT treatment (modality conversion) will be recorded and reported. Treatment breaks and delays due to dosimetric concerns, replans or change in modalities will be recorded.
Comparison of planned versus delivered dose for PBT plans | From date of first patient enrolment until the date of the last patient treatment (up to 36 months)
  Compare planned dose versus estimated delivered dose, calculated with review of daily online imaging, for PBT plans.
Local control at 2 years | 2 years from the end of recruitment
  Local control at 2 years as assessed clinically.
Event free survival and overall survival at 2 years | 2 years from the end of recruitment
  Event free survival and overall survival at 2 years assessed clinically.
Acute toxicity and late toxicity | 6 weeks after the end of treatment
  Acute toxicity measured by clinician assessment and patient reported outcome questionnaire. Late toxicity measured by clinician assessment.

IPD SHARING:
Plan to Share IPD: Undecided